CLINICAL TRIAL: NCT02506374
Title: Project BEST-Sleep: A Pilot Study to Develop a Biobehavioral Self-Management Therapeutic Intervention for Sleep in Alzheimer/Caregiver Dyads
Brief Title: Development of Therapeutic Intervention for Sleep in Alzheimer/Caregiver Dyads
Acronym: BEST-Sleep
Status: Withdrawn | Type: Observational
Why Stopped: Never able to get any subjects enrolled
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1412015088
Record Dates: First submitted 2015-07-16; First posted 2015-07-23 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
This non-intervention qualitative study will use focus groups to assess the feasibility and acceptability of a proposed intervention for a future study. The focus group will discuss a potential biobehavioral family self-management intervention designed to improve sleep in persons with Alzheimer's disease (PAD) and their caregivers (CG).

DETAILED DESCRIPTION:
Approximately 16 caregivers of home-based PAD/CG dyads (person with Alzheimer's disease/caregiver dyads) will be recruited from the community. A series of two audiotaped focus groups will be conducted with these caregiver participants. The first focus group will explore perspectives on what constitutes a feasible and acceptable intervention to improve their sleep and associated symptoms. The second focus group will consist of follow up and confirmation of findings from the first focus group. The intervention will be developed and refined based upon focus group findings.

ELIGIBILITY:
Inclusion Criteria:

1. screen positive on the PROMIS sleep disturbance and associated symptoms measures
2. be a caregiver within a PAD/CG dyad
3. speak/understand English
4. agree to be audiotaped during focus group participation
5. be at least 18 years of age

Exclusion:

1. they negative on the PROMIS sleep disturbance and associated symptoms measures,
2. are not a caregiver within a PAD/CG dyad,
3. do not speak/understand English,
4. refuse to take part in audiotaping of the focus groups,
5. are not at least 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers of home-based PAD/CG dyads (person with Alzheimer's disease/caregiver dyads) will be recruited from the community
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Qualitative Output from Focus Groups | 1 day
  Focus group data will be processed utilizing Atlas.ti software and analyzed using the constant comparative method.

CONTACTS AND LOCATIONS:
Overall Officials: LuAnn Etcher, PhD, Principal Investigator — Yale University
Locations (1):
- Jewish Senior Services, Fairfield, Connecticut, United States